CLINICAL TRIAL: NCT01186237
Title: Early Removal of Urinary Catheters in Patients After Rectal Surgery: a Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REC0004; SU-05272010-6187 (Other: Stanford University); 17865 (Other: Stanford University); NCI-2010-02350
Record Dates: First submitted 2010-08-09; First posted 2010-08-23 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Colorectal Cancer
Keywords: Colon/Rectal Cancer Rectal Cancer; Quality of Life
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Early urinary catheter removal (Experimental)
  Interventions: Procedure: Early urinary catheter removal

INTERVENTIONS:
Procedure: Early urinary catheter removal — All patients will have foley catheters removed between 0600 and midnight of post-operative day 3 (Day 0 being the day of operation).

SUMMARY:
Recent national surgical quality guidelines (Surgical Care Improvement Project, National Hospital Inpatient Quality Measures)state that removal of urinary catheters should occur by post-operative day two for all surgical patients. These guidelines exclude neither patients who have undergone rectal surgery nor those with epidural analgesic catheters. The common practice among most colorectal surgeons is to leave urinary catheters in for three to five days for patients who have undergone rectal operations, due to concern for urinary retention. This study aims to explore the outcomes of following the national surgical guidelines for early urinary catheter removal, especially with regards to urinary retention and urinary tract infection.

DETAILED DESCRIPTION:
All patients undergoing anterior resection (rectosigmoid), low anterior resection, abdomino-perineal resection, total proctocolectomy with ileal pouch-anal anastomosis, sigmoid colectomy, and coloanal anastomosis will be included in the study. All patients will undergo standard pre-operative work-up prior to the operation. As part of the operative note, the level of the anastomosis must be documented.

1. All patients will have foley catheters removed between 0600 and midnight of post-operative day 3 (Day 0 being the day of operation).
2. All patients will undergo bladder ultrasound prior to catheter removal.
3. All patients will undergo bladder ultrasound by nursing staff six hours after catheter removal, and after voiding the first time after catheter removal, or if the patient experiences symptoms of urinary retention.

6. Patients who meet definition of urinary retention (>100cc post-void residual) will undergo intermittent straight catheterization every six hours or with symptoms. For those who refuse intermittent straight catheterization, a indwelling urinary catheter will be inserted and left in for 24 hours before removal.

7. For patients who have low urine output indicating under-resuscitation, indwelling catheters will be re-inserted and removed when ongoing resuscitation measures are completed.

8. For patients who are actively undergoing fluid resuscitation on post-operative day 3 will not have their urinary catheters removed until resuscitation and monitoring is complete.

9. Patients who report symptoms of benign prostatic hypertrophy (BPH) and/or are already on medications for BPH will be continued on those medications starting on post-operative day 1.

10. Patients who have persistent urinary retention when they are otherwise ready to be discharged home will be sent home with a leg bag and follow up in urology clinic for voiding trial in 1-2 weeks.

11. Urinalysis/urine culture will be performed for symptomatic patients.

ELIGIBILITY:
Inclusion criteria

All patients at Stanford Hospital undergoing:

* anterior resection
* sigmoid colectomy
* low anterior resection
* abdomino-perineal resection
* total proctocolectomy with ileal pouch-analanastomosis
* coloanalanastomosis.

Exclusion criteria Patients with history of neurogenic bladder who had indwelling catheters or required intermittent straight catheterization prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
urinary retention | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lane Welton, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States